CLINICAL TRIAL: NCT06642298
Title: Studying the Impact of Religiosity/Spirituality on the Severity of Depression and Anxiety in Patients Attending Psychiatry Unit of Assiut University Hospitals
Brief Title: Studying Impact of Religiosity and Spirituality on Depression and Anxiety
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Ahmed Abdelrahman Ali, Principal Investigator, Assiut University
Other Study IDs: RSDAP
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Depression; Anxiety
Keywords: Depression; Anxiety; Religiosity; Spirituality; Egypt
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to detect correlation between religiosity/spirituality and severity of depression and anxiety as well as finding impact on quality of life in patients, suffering from one of those disorders or both, who are attending the Psychiatric Clinic and Ward of Assiut University Hospitals. Given the centrality of religious activities in Egyptian society and the Arab population as a whole, finding such correlation may be beneficial in terms of analysing factors that may lead to depression and/or anxiety as well as factors that may reduce their severities.

DETAILED DESCRIPTION:
Religiosity and spirituality are fundamental aspects of the human experience, shaping beliefs, values, and how individuals navigate life's challenges. Religiosity refers to the degree to which individuals identify with, and participate in the practices and beliefs of, a particular religion. It encompasses behaviors like prayer, attending religious services, and following religious teachings. Spirituality, on the other hand, is a broader concept that reflects a sense of connection to something larger than oneself, a search for meaning and purpose in life. This connection can be expressed through religious beliefs, but it can also be independent of religion, encompassing a connection to nature, humanity, or a sense of purpose. Research has increasingly explored the complex interplay between these constructs and mental health. The relationship between religiosity/spirituality and mental health is multifaceted. Religious involvement can provide individuals with social support, a sense of belonging, and a framework for coping with stress. Spiritual beliefs can offer comfort, hope, and a sense of purpose, potentially promoting resilience in the face of challenges. However, the relationship is not always straightforward. Certain religious beliefs or practices could contribute to feelings of guilt, shame, or isolation, potentially impacting mental health. Additionally, negative religious coping styles, such as feeling angry or abandoned by God, might exacerbate mental health problems. Given the centrality of religion in the Arab world, including Egypt, a deeper look into the associations between religiosity/spirituality and psychiatric disorders such as depression and anxiety is warranted.

ELIGIBILITY:
* Inclusion Criteria:

  1. Age above 18 years old.
  2. Diagnosed with Depression and/or Anxiety disorders according to the DSM-5 criteria.
* Exclusion Criteria:

  1. Severe psychiatric disorders including schizophrenia, personality disorders and drug-use disorders.
  2. Patients with cognitive impairment.
  3. Severe comorbid medical condition or disabilities including metabolic diseases and neurological disabilities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 diagnosed with depression and/or anxiety who attend the Psychiatry hospital in Assiut University.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between religiosity/spirituality and severity of depression and/or anxiety. | 2 years
  Correlation between religiosity/spirituality and severity of depression and/or anxiety. Religiosity/Spirituality measures will include Centrality of Religiosity 5 and the Spiritual Well-Being Scale. Depression and Anxiety severity will be assessed by Hamilton Scale.

SECONDARY OUTCOMES:
Quality of Life by WHOQOL-BREF Scale score | 2 years
  Assessing quality of life by using the The WHO Quality of Life (WHOQOL - BREF) scale, which is a widely used tool for assessing an individual's perceived quality of life across various domains. The Arabic version of this scale is designed to measure the quality of life in Arabic-speaking populations, considering cultural and linguistic differences.

REFERENCES:
- [Background] Hill PC, Hood RW. Measures of Religiosity. Birmingham: Religious Education Press; 1999
- [Background] Miller WR, Thoresen CE. Spirituality and Health: What We Know, What We Need to Know. Journal of Behavioral Medicine. 2003;26(1):1-11
- [Background] Pargament KI. The Psychology of Religion and Coping: Theory, Research, Practice. New York: Guilford Press; 1997.
- [Background] First MB, Spitzer RL, Gibbon M, Williams JBW. Structured Clinical Interview for DSM-IV Axis I Disorders (SCIDI), Clinician Version. New York: New York Psychiatric Institute; 1997
- [Background] Hamilton M. Development of a rating scale for primary depressive illness. Br J Soc Clin Psychol. 1967 Dec;6(4):278-96. doi: 10.1111/j.2044-8260.1967.tb00530.x. No abstract available. PMID 6080235
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] Huber S, Huber OW. The Centrality of Religiosity Scale (CRS). Religions. 2012;3(3):710-724
- [Background] Paloutzian RF, Ellison CW. Loneliness, spiritual well-being, and the quality of life. In: K. S. Schaefer & S. S. M. Cohen, editors. Measurement of Meaningful Life. New York: Wiley; 1982. p. 222-233
- [Background] The World Health Organization Quality of Life Assessment (WHOQOL): development and general psychometric properties. Soc Sci Med. 1998 Jun;46(12):1569-85. doi: 10.1016/s0277-9536(98)00009-4. PMID 9672396